CLINICAL TRIAL: NCT05798156
Title: A Prospective Multicenter Phase 2 Study of the Chemotherapy-light Combination of Intravenous Rituximab With the Antibody-drug Conjugate Polatuzumab Vedotin and the Bispecific Antibody Glofitamab in Previously Untreated Aggressive B-cell Lymphoma Patients Above 60 Years of Age Ineligible for a Fully Dosed R-CHOP
Brief Title: Rituximab in Combination With Glofitamab and Polatuzumab Vedotin in Patients With Previously Untreated Aggressive B-cell Lymphoma Ineligible for R-CHOP
Acronym: R-Pola-Glo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Salzburg (Other); Arbeitsgemeinschaft medikamentoese Tumortherapie (Other); Roche Pharma AG (Industry); Zentrum für Klinische Studien Leipzig (Other); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-Pola-Glo; ML44400 (Other Grant/Funding Number: Roche); 2022-003398-51 (EudraCT Number); GLA 2022-10 (Other: GLA); NHL-16 (Other: AGMT); IKF-t062 (Other: Frankfurter Institut für klinische Krebsforschung IKF GmbH)
Record Dates: First submitted 2023-03-08; First posted 2023-04-04 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab; Rituximab; obinutuzumab; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- chemolight R-Pola-Glo treatment (Experimental)
  Interventions: Drug: Glofitamab; Drug: Rituximab; Drug: Obinutuzumab; Drug: Polatuzumab vedotin

INTERVENTIONS:
Drug: Glofitamab — Glofitamab is a fully humanized, engineered monoclonal bivalent antibody of the IgG1 isotype.
Drug: Rituximab — Rituximab is a genetically engineered chimeric mouse/human anti-CD20 monoclonal antibody
Drug: Obinutuzumab — Obinutuzumab is a fully humanized, glycoengineered type II monoclonal antibody of the IgG1 isotype that binds to an epitope on CD20
Drug: Polatuzumab vedotin — Polatuzumab vedotin is an antibody-drug-conjugate that contains a humanized IgG1 anti-CD79b monoclonal antibody (MCDS4409A) and a potent anti-mitotic agent (MMAE) linked through a protease-cleavable linker.

SUMMARY:
In the present trial the chemotherapy- light treatment concept R-Pola-Glo will be evaluated that combines the anti-CD20 antibody rituximab (R) with the ADC polatuzumab vedotin (Pola) and the (BiMabs) glofitamab (Glo) in elderly and/or medical unfit and previously untreated patients with aggressive B-cell lymphoma. The outcome and feasibility data obtained here will be used for further clinical development of this new chemolight triple combination.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent and is able and willing to comply with the study protocol and protocol mandated treatments according to ICH and local regulations.
2. Patient is above 60 years of age
3. Patient is not eligible for a fully dosed R-CHOP
4. Patient has histologically confirmed aggressive B-cell lymphoma.
5. Patient has at least one measurable FDG PET-positive lymphoma manifestation; defined as lesional maximum FDG uptake higher than the maximum FDG uptake in unaffected liver parenchyma as measured in a reference volume-of-interest with >10 mL
6. Baseline biopsy material is available for central review.
7. Female patients considered as women of childbearing potential (WOCBP, see section 5.2.7 for definition) and male patients with female partners considered as WOCBP must:

   1. agree to either remain completely abstinent (refrain from heterosexual intercourse) or to use at least one effective contraceptive methods that results in a failure rate of < 1% per year
   2. refrain from donating ova (female patients) or donating sperm (male patients)
   3. in case of male patients with pregnant female partners, remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures such as a condom to avoid exposing the embryo.
8. Patient did not receive any prior systemic lymphoma therapy.
9. Patient has an ECOG performance status of ≤ 2.
10. Patient has with treatment a life expectancy (in the opinion of the investigator) of at least 12 weeks.
11. Patient has adequate liver function
12. Patient as adequate hematological function
13. Patient has adequate renal function
14. Patients has negative serologic and/or polymerase chain reaction (PCR) test results for:

    * Acute or chronic hepatitis B (HBV) infection.
    * Hepatis C virus (HCV) and human immunodeficiency virus (HIV)
15. Patient has no active SARS-CoV-2 infection.

Exclusion Criteria:

Medical conditions:

1. Patient with chronic lymphocytic leukemia (CLL), acute lymphoblastic leukemia (ALL) (including CD20+ ALL), lymphoblastic lymphoma, Richter's transformation, Burkitt lymphoma.
2. Patient ≤ 60 years
3. Patient with known active infection, or reactivation of a latent infection, whether bacterial (e.g., tuberculosis), viral (including, but not limited to severe pneumonia, COVID-19, Epstein-Barr virus [EBV], cytomegalovirus [CMV], hepatitis B, hepatitis C, and HIV], fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 4 weeks prior to study enrollment.
4. Patient with current > Grade 1 peripheral neuropathy.
5. Patient with history of confirmed progressive multifocal leukoencephalopathy (PML).
6. Patient with history of leptomeningeal disease.
7. Patient with current or history of CNS lymphoma.
8. Patient with current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease with exceptions.
9. Patient with another invasive malignancy in the last 2 years (with the exception of basal cell carcinoma and tumors deemed by the Investigator to be of low likelihood for recurrence), with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate 90%), such as adequately-treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
10. Patient with significant or extensive history of cardiovascular disease (such as New York Heart Association (NYHA) Class ≥ II cardiac disease, congestive heart failure, myocardial infarction or cerebrovascular accident within the past 3 months, unstable arrhythmias, or unstable angina or history of multiple cardiovascular events) or significant pulmonary disease (including obstructive pulmonary disease and history of bronchospasm).
11. Patient with active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis (see addendum for a more comprehensive list of autoimmune diseases and immune deficiencies), with exceptions.
12. Patient with uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).
13. Patient with history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic.

    Prior/Concomitant Therapy:
14. Patient received treatment with any other standard anti-cancer radiotherapy/chemotherapy including investigational therapy (defined as treatment for which there is currently no regulatory authority approved indication) within 4 weeks or five times the elimination half-life of the product, whichever is longer, prior to study enrollment.
15. Patient with prior solid organ transplantation.
16. Patient with prior allogeneic stem cell transplantation.
17. Patient with prior treatment with targeted therapies (e.g., tyrosine kinase inhibitors, systemic immunotherapeutic/immunostimulating agents, including, but not limited to, CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies, radio-immunoconjugates, antibody-drug conjugates, immune/cytokines, and monoclonal antibodies) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to study enrollment.
18. Patient with toxicities from prior anti-cancer therapy including immunotherapy that did not resolve to ≤ Grade 1 except for alopecia, endocrinopathy managed with replacement therapy and stable vitiligo.
19. Patient with any history of immune related ≥ Grade 3 AE except for endocrinopathy managed with replacement therapy.
20. Patient with ongoing corticosteroid use 25 mg/day of prednisone or equivalent within 4 weeks prior and during study treatment.
21. Patient with treatment with systemic immunosuppressive medication (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with exceptions.
22. Patient who received administration of a live, attenuated vaccine within 4 weeks prior to study enrollment infusion or anticipation that such a live, attenuated vaccine will be required during the study or within 5 months after the last dose of study treatment.

    Other Exclusions:
23. Patient with history of illicit drug or alcohol abuse within 12 months prior to screening, in the Investigator's judgment.
24. Patient with history of severe allergic anaphylactic reactions to chimeric or humanized monoclonal antibodies or recombinant antibody-related fusion proteins.
25. Patient with known hypersensitivity to Chinese hamster ovary (CHO) cell products or to any component of the rituximab, obinutuzumab, polatuzumab vedotin and/or glofitamab formulation and/or to the contrast agents used in the study.
26. Female patient is pregnant or breast feeding. Female patients of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment.
27. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.
28. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts.
29. Patients who are dependent on the sponsor, the investigator or the trial site.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
1 year progression-free survival (PFS) rate of the first 80 patients | 12 months
  defined as the time from the day of inclusion until disease progression (PD) or relapse after complete remission (CR), or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Event-free survival (EFS) | 54 months
  defined as the time from the day of inclusion until progressive disease or relapse after complete remission, initiation of subsequent systemic antilymphoma treatment, radiation of single PET-CT positive lesions or death due to any cause, whichever occurs first.
Overall survival (OS) | 54 months
  defined as the time from the day of inclusion until death due to any cause
Response rate at different timepoints | 6 weeks, 18 weeks, 36 weeks
  Response rates after 2 cycles (during target dose phase), 6 cycles (end of target dose phase before start of consolidation phase) and 12 cycles (end of treatment following completion of consolidation phase). i.e., complete remission (CR) rate, partial remission (PR) rate, overall remission rate (ORR: CR+PR), stable disease (SD) rate and progressive disease (PD) rate
Relapse rate | 54 months
  defined as the number of patients with relapse, divided by the number of patients achieving C
Conversion rate of PR to CR | 54 months
  defined as the number of patients achieving mCR at the end of study treatment (including consolidation phase) divided by the number of patients achieving PR after end of target dose phase (before start of consolidation phase)
Duration of response (DoR) | 54 months
  defined as the time from documentation of CR until relapse or lymphoma associated death without documented relapse
Rate and type of adverse events (AEs) and serious adverse events (SAEs) | 54 months
Rate of secondary malignancies | 54 months
  defined as the number of patients with secondary malignancies divided by the number of analyzable patients
Treatment-related death rate | 54 months
  defined as the number of treatment related deaths during therapy or up to 2 months after the end of study treatment, but before the start of further treatment, divided by the number of analyzable patients
Protocol adherence | 54 months
  number and duration of R-Pola-Glo cycles, number and duration of glofitamab maintenance, cumulative and relative doses of rituximab, glofitamab and polatuzumab.
Patient-reported outcomes for quality of life (QoL): EORTC QLQ-C30 | 54 months
  measured by EORTC QLQ-C30 (a 30-item questionnaire developed by the European Organisation for Research and Treatment of Cancer). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Patient-reported outcomes for quality of life (QoL): FACT-Lym | 54 months
  measured by FACT-Lym (Functional Assessment of Cancer Therapy - Lymphoma; scores from 0 - 4; The higher the score, the better the QOL)

OTHER OUTCOMES:
Rate of minimal residual disease (MRD)-negative patients after end of target phase and at end of treatment | 54 months
Duration of molecular remission for MRD negative patients | 54 months
Outpatient setting w/o hospitalization | During Cycle 1-6
  Proportion of patients in whom R-Pola-Glo medication can be administered in the outpatient setting as recommended by the safety board (judged before treatment and including modification after cycle 1 or 2) and no hospitalization occurs following 24hrs after last administration.
Outpatient setting with hospitalization | During Cycle 1-6
  Proportion of patients in whom R-Pola-Glo medication can be administered in the outpatient setting as recommended by the safety board (judged before treatment and including modification after cycle 1 or 2) but are hospitalized within 24hrs after last administration for timely medical assistance from treating physician for symptoms developed following treatment with R-Pola-Glo.
Cycles safely administered in outpatient setting per patient. | During Cycle 1-12

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Institut fuer Klinische Krebsforschung IKF GmbH
Locations (30):
- Austria (8):
  - Uniklinik Innsbruck, Innsbruck
  - Kepler Universitätsklinikum, Linz
  - Ordensklinikum Linz - Barmherzige Schwestern, Linz
  - Ordensklinikum Linz - Elisabethinen, Linz
  - Landeskrankenhaus Salzburg Universitätsklinikum der Paracelsus Medizinischen Privatuniversität, Salzburg
  - Univ. Klinikum St. Pölten, Sankt Pölten
  - AKH Meduni Wien, Vienna
  - Hanusch Krankenhaus, Vienna
- Germany (22):
  - Universitätsklinikum Magdeburg, Magdeburg, Saxony-Anhalt
  - Charité - Universitätsmedizin Berlin, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Medizinisches Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Klinikum Chemnitz, Chemnitz
  - Uniklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Ev. Klinikum Essen-Mitte, Essen
  - Westdeutsches Tumorzentrum Essen, Essen
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Halle, Halle
  - University Hospital Jena, Jena
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Leverkusen, Leverkusen
  - Klinikum Ludwigshafen, Ludwigshafen
  - TU München (rechts des Isar), München
  - Unversitätsklinikum Münster, Münster
  - Ortenauklinikum Offenburg-Kehl, Offenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Kreiskliniken Reutlingen, Reutlingen
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.